CLINICAL TRIAL: NCT01753635
Title: Comparison of the Baska Mask Airway to a Single-use LMA Device in Low-risk Female Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: John Laffey (Other)
Responsible Party: Sponsor-Investigator, John Laffey, Professor of Anaesthesia and Critical Care, Consultant Anaesthetist, University College Hospital Galway
Organization: University College Hospital Galway (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C.A.724
Record Dates: First submitted 2012-12-17; First posted 2012-12-20 (Estimated); Last update posted 2013-03-19 (Estimated); Status verified 2013-03

CONDITIONS: Performance and Safety of an Airway Management Device
Keywords: Baska mask; LMA; single use LMA device; laryngeal mask airway; supraglottic airway device

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Baska mask (Experimental): In this arm the Baska mask will be used as the airway management device
  Interventions: Device: supraglottic airway placement and use
- single use laryngeal mask airway device (LMA) (Active Comparator): in this arm a single use LMA device will be used for airway management.
  Interventions: Device: supraglottic airway placement and use

INTERVENTIONS:
Device: supraglottic airway placement and use

SUMMARY:
The purpose of this study is to compare the performance of the Baska mask supraglottic airway device with a single use laryngeal mask device (LMA) in low-risk female patients.

The investigators have performed a number of studies on novel airway devices, including 3 studies on the Baska mask. This trial will compare some performance characteristics of the studied devices, including airway seal pressures, insertion success rates, device use difficulty scores. Additional performance and device safety data will be accumulated.

The investigators have two primary hypotheses, namely 1.Non-inferiority of first placement attempt success rate of the Baska mask vs LMA; and 2.greater seal pressure of the Baska mask vs LMA.

DETAILED DESCRIPTION:
Supraglottic airway devices have established place in the airway management in patients undergoing general anesthesia.

The Baska mask is a new supraglottic airway device. It's features include:

1. Non pressurized cuff designed to reduce the risk of oropharyngeal tissue damage.
2. Improved cuff seal during the inspiratory phase of positive pressure ventilation
3. An improved system for drainage of oropharyngeal contents intended to reduce the rate of lung aspiration.
4. Integrated bite-block to reduce the risk of patients biting and blocking the airway.

This study is randomized, single-blinded, controlled trial. The participants will be allocated to two groups, in which either the Baska mask or the single use LMA will be the primary airway management device.

Clinical Research Ethics Committee approval has been obtained. Suitable participants will be recruited after written informed consent.

Standard anesthetic preassesment and anesthesia will be provided.

Consenting patients will be randomly allocated to either of the 2 study groups.

Protocol for airway size selection and attempts at placement will be followed.

The investigators will monitor a number of parameters, including time and ease of insertion, airway seal pressure, airway leak, complications related to device use and other.

Follow up will be performed.

The investigators have two primary hypotheses:

1. That the Baska mask is non-inferior to LMA in respect if first placement attempt success rate. A greater than 15% difference in success rate will be considered a clinically important difference and will disprove this hypothesis.
2. The Baska mask is superior in respect of seal pressure. A 20% higher seal pressure with Baska as compared to the LMA device seal pressure will be considered a clinically important difference.

Interim analysis will be performed once 75 patients are recruited per group. This is reasonable as this figure exceeds that required to prove or disprove the primary hypothesis regarding the seal pressure. The study will only be stopped at this stage if the non-inferiority hypothesis is disproven with P value < 0.01

In addition to the above the investigators will evaluate a number of secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Written informed consent
* ASA 1-3
* No relevant allergies
* Body-mass index (BMI) 35 or less
* Age 16-85
* Non-urgent surgery of planned duration under 4 hours

Exclusion Criteria:

* Inability of patient/parent to understand or consent for the trial
* Neck pathology
* Previous or anticipated problems with the upper airway or upper GI tract
* BMI >35
* Predicted or previously documented difficult airway
* Live Pregnancy
* Increased risk for Gastric Aspiration

Ages: 16 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2012-11; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Rate of successful placement of the supraglottic device on first attempt | within 30 minutes of commencement of general anesthesia
  The hypothesis is that the Baska mask will have first time placement attempt success rate that is no more than 15% less than that of the comparator - a single use LMA device.
Seal pressure of the supraglottic device | Within 30 minutes of commencement of general anesthesia
  The investigators will measure the airway seal provided by the device used. The hypothesis is that the seal pressure of the Baska mask is 20% higher than that of the comparator single-use LMA device.

SECONDARY OUTCOMES:
Overall rate of successful placement of the supraglottic device | Within 30 minutes of commencement of general anesthesia. Up to 3 device placement attempts are allowed.
Number of device placement attempts | Within 30 minutes of commencement of general anesthesia
Number of optimization maneuvers during device placement | Within 30 minutes of commencement of general anesthesia
user rated Device difficulty score | within 30 minutes of commencement of general anesthesia
  the investigators will use 10 cm visual analogue scale to score the whole experience of using the device until successful ventilation is achieved.
vitals parameter stability | in the period immediately before and within the first 35 minutes of general anesthesia
  The investigators will record non-invasive arterial oxygen saturation, heart rate and blood pressure preoperatively, after induction of general anesthesia and after placement of the airway device.
Laryngeal view obtained on fiberoptic assessment | within 2 hours of commencement of general anesthesia
  The investigators will perform this when feasible.
Complication rates | from the moment general anesthesia commenced up to 3 days postoperatively
  Complications specifically monitored will be: blood staining, laryngospasm, lip damage, throat pain, dysphagia, dysphonia, heartburn, nausea and vomiting.
  The investigators will record other complications related to the use of the device, including but not limited to: desaturation, need to reposition device or switch to alternative device, teeth damage, regurgitation, aspiration

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Neligan, FFARCSI, Principal Investigator — Galway University Hospitals
Locations (1):
- Galway University Hospitals, Galway, Ireland